CLINICAL TRIAL: NCT01345851
Title: Image-Guided Hypofractionated Radiotherapy With Stereotactic Boost and Chemotherapy for Inoperable Stage II-III Non-Small Cell Lung Cancer
Brief Title: Image-Guided Hypofractionated Radiation Therapy With Stereotactic Body Radiation Therapy Boost and Combination Chemotherapy in Treating Patients With Stage II-III Non-Small Cell Lung Cancer That Cannot Be Removed By Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-001342; NCI-2011-00673 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-04-27; First posted 2011-05-02 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Large Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Image-Guided; Carboplatin; Paclitaxel; Taxes; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dose-escalation of RT) (Experimental): Patients undergo image-guided hypofractionated RT over 35 minutes 5 days a week for 2 weeks followed by 5 fractions of hypofractionated RT boost. Patients also receive standard carboplatin and paclitaxel for 3 weeks.
  Interventions: Radiation: hypofractionated radiation therapy; Other: laboratory biomarker analysis; Radiation: image-guided radiation therapy; Drug: carboplatin; Drug: paclitaxel; Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Radiation: hypofractionated radiation therapy — Undergo image-guided hypofractionated Radiation Therapy over 35 minutes 5 days a week for 2 weeks
Other: laboratory biomarker analysis — Correlative studies
Radiation: image-guided radiation therapy — Undergo 5 fractions of image-guided hypofractionated Radiation Therapy boost.
Drug: carboplatin — The maximal chemotherapy treatment dose for carboplatin during the 3 week radiation therapy is AUC 2.
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel — The maximal chemotherapy treatment dose for paclitaxel during the 3 week radiation therapy is 45mg/m2.
  Other Names: Anzatax; Asotax; TAX; Taxol
Radiation: stereotactic body radiation therapy — Undergo hypofractionated RT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy

SUMMARY:
This clinical trial studies image-guided hypofractionated radiation therapy (RT) when given together with hypofractionated RT boost and combination chemotherapy in treating patients with stage II-III non-small cell lung cancer (NSCLC) that cannot be removed by surgery. RT uses high energy x-rays to kill tumor cells. Hypofractionated RT may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving RT together with combination chemotherapy may kill more tumor cells and allow doctors to save the part of the body where the cancer started

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) using hypofractionated RT in patients with stage II-III NSCLC.

SECONDARY OBJECTIVES:

I. To determine the dose-limiting toxicity, if the MTD is reached.

II. To determine the tumor local control (LC).

III. To determine the lung cancer disease specific survival (DSS).

IV. To determine the overall survival (OS).

V. To assess the transforming growth factor-beta (TGF-B), interleukin (IL)-1, and IL-6 levels as predictive biomarkers for treatment induced tissue injury.

OUTLINE: This is a dose-escalation study of image-guided hypofractionated RT.

Patients undergo image-guided hypofractionated RT over 35 minutes 5 days a week for 2 weeks followed by 5 fractions of hypofractionated RT boost. Patients also receive standard carboplatin and paclitaxel for 3 weeks.

After completion of study treatment, patients are followed up at 4-6 weeks, every 3 months for the first 2 years, and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary non-metastatic NSCLC; eligible histological subtypes include: squamous cell carcinoma, adenocarcinoma, squamous-adeno carcinoma, large-cell carcinoma, and non-small cell carcinoma not otherwise specified
* Clinical stage II and III NSCLC as defined by American Joint Committee on Cancer (AJCC) Cancer Staging Manual, seventh edition; acceptable imaging modalities to document nodal positivity include computed tomography (CT) chest, positron emission tomography (PET)-CT, or thoracic magnetic resonance imaging (MRI)
* For clinically stage II patients, the patient must have been evaluated by a thoracic surgeon, and deemed medically or technically inoperable, or the patient must refuse surgery
* Karnofsky performance status >= 70
* If a woman is of childbearing potential, a negative serum pregnancy test must be documented; women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) for duration of study treatment and for up to 4 weeks following the study treatment

Exclusion Criteria:

* Patients who have previously received therapeutic radiation therapy to the chest
* Active systemic, pulmonary, or pericardial infection
* Use of concurrent gemcitabine-based chemotherapy during radiotherapy
* Pregnant women, or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception for the entire study period and for up to 4 weeks after the study treatment
* Refusal to sign the informed consent
* Patients who are participating in a concurrent treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-03-23 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To determine the maximal tolerated dose using hypofractionated radiotherapy in patients with stage II-III non small cell lung cancer. | up to 90 days
  The primary end point is to reach the maximum tolerated dose or a total of 75 Gy, whichever comes first, by escalating the daily dose of last 5 fractions.

SECONDARY OUTCOMES:
To determine tumor Local control | participants will be followed for 2 years
  Radiological evaluation (CT, PET-CT) will be done to assess tumor.
To determine Lung cancer Disease specific survival | Participants will be followed for 2 years
Overall survival | Participants will be followed for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Percy Lee, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Wu TC, Luterstein E, Neilsen BK, Goldman JW, Garon EB, Lee JM, Felix C, Cao M, Tenn SE, Low DA, Kupelian PA, Steinberg ML, Lee P. Accelerated Hypofractionated Chemoradiation Followed by Stereotactic Ablative Radiotherapy Boost for Locally Advanced, Unresectable Non-Small Cell Lung Cancer: A Nonrandomized Controlled Trial. JAMA Oncol. 2024 Mar 1;10(3):352-359. doi: 10.1001/jamaoncol.2023.6033. PMID 38206614